CLINICAL TRIAL: NCT00977184
Title: Controlled Study of 50 Hz Repetitive Transcranial Magnetic Stimulation for the Treatment of Parkinson's Disease
Brief Title: 50 Hz Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Mark Hallett, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 090221; 09-N-0221
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Transcranial Magnetic Stimulation (TMS); Treatment Study; PD; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Experimental)
  Interventions: Procedure: 50 HZ Repetitive TMS
- Sham rTMS (Sham Comparator)
  Interventions: Procedure: Sham rTMS

INTERVENTIONS:
Procedure: 50 HZ Repetitive TMS
  Arms: Real rTMS
Procedure: Sham rTMS
  Arms: Sham rTMS

SUMMARY:
Background:

* In transcranial magnetic stimulation (TMS), a device creates a short-lasting magnetic field which induces an electric current in the brain leading to a change in the activity of brain cells. There are different effects on the brain with different rates of stimulation. In a previous study in people with Parkinson's disease, repetitive TMS (rTMS) given at a particular rate temporarily improved their ability to walk. A faster rate of rTMS may be more effective in treating symptoms than the rate originally used.
* This study will compare active rTMS to inactive (sham or Placebo) rTMS. Half of the people in this study will have active rTMS; the other half will have no brain stimulation with rTMS.

Objectives:

- To see if a faster rate of transcranial magnetic stimulation is a more effective treatment for the symptoms of Parkinson's disease than the slower rates that have been studied.

Eligibility:

* Individuals between 40 and 80 years of age who have been diagnosed with mild or moderate Parkinson's disease.
* Participants must currently be taking Sinemet or dopamine agonists drugs (e.g., bromocriptine, cabergoline, pergolide, pramipexole, ropinirole, apomorophine, and rotigotine), and are willing to continue their same treatments for the duration of the study.

Design:

* This study requires 11 outpatient visits to the NIH Clinical Center over 6 weeks. Participants can also be admitted and stay as an inpatient in the NIH Clinical Center for the entire study period (for the 10 visits during the first weeks and the follow-up visit a month later).
* Initial visit will consist of a physical examination; a test of participants' time to walk 10 meters; and questions about memory, mood, and quality of life. Participants should not take Parkinson's disease medications for 12 hours before this visit; once the examinations and tests are complete, participants will be able to take the medications. Researchers will repeat the tests 1 hour after participants take the medication.
* TMS sessions: 8 TMS sessions (4 sessions per week) over 2 weeks. Each stimulation session will last half an hour. Half of the participants will receive active TMS; the other half will receive sham TMS.
* The first 10 participants will have additional tests to study the safety of rapid TMS in patients with Parkinson's disease.
* A day after completing the last TMS session, participants will repeat the same tests as the first visit before and after taking their medication as in the first assessment and respond to questions about mood, memory, and quality of life.
* One month after completing the last TMS session, participants will repeat the same tests as the first visit before and after taking their medication.

DETAILED DESCRIPTION:
Objective:

To demonstrate cumulative and long-lasting improvement of parkinsonian symptoms by 50 Hz rTMS (repetitive transcranial magnetic stimulation) and its safety in Parkinson's Disease (PD) patients.

Study population:

Up to 30 PD patients in Hoehn and Yahr disease stage 2-4 while off medication will be enrolled. Patients must be receiving more than 300 mg of levodopa (including dopamine agonists) and have gait problems.

Design:

This is a randomized, double-blind, placebo (sham)-controlled study of 26 patients with PD in 2 groups (real versus sham stimulation). The study involves performance (8 interventions) of 50 Hz rTMS with large circular coil over the motor cortex on both sides of the brain. Assessment of PD symptoms with standard tests of motor function will be performed over a one-month period.

Outcome measure:

The primary endpoint include the changes in gait speed as assessed by the time it takes to walk 10 meters and the changes in bradykinesia as assessed by measuring the time it takes to do 10 combined hand and arm movements.

Secondary endpoints include the changes in the total, motor and activities of daily living Unified Parkinson's Disease Rating Scale (UPDRS) score.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women aged 40 to 80 years with DOPA-responsive PD

Hoehn and Yahr grade of 2 to 4 while off

Must be on a regimen including levodopa

Total dose of levodopa and dopamine agonists (using dopamine equivalents) has to be equal to or more than 300 milligrams per day

problems with walking and gait time for a 10-meter distance greater than six seconds or more

EXCLUSION CRITERIA:

Any active psychiatric disease

History of seizures and epilepsy

Concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drugs other than anti-parkinsonian agents that could lower the seizure threshold except for SSRI

Pallidotomy, implanted electrodes and generator for deep brain stimulation

Pregnancy

Surgically or traumatically implanted foreign bodies such as a pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during TEP.

Study would cause undue risk or stress for reasons such as tendency to fall, excessive fatigue, general frailty, or excessive apprehensiveness.

Dementia as assessed by the Folstein's Mini-Mental Test Examination (MMSE less than or equal to 24/30) or mentally impaired patients having no capacity to provide their own consent (the physician establishing the diagnosis and applying UPDRS will evaluate patient's mental capacity using conventional clinical interview)

Unable to walk a 10-meter distance.

More than occasional falls, i.e. daily falls (corresponding to a score greater than or equal to 3 and more in UPDRS item 13), history of fall(s) with significant injuries, absence of postural response in the on and/or spontaneous loss of balance in the off condition (corresponding to a score of greater than or equal to 2 and greater than or equal to 3 in on/off condition, respectively, in UPDRS item 30)

Pregnancy is unusual in patients with PD, grade 2-4. Urine sample for the pregnancy test will be obtained in patients of childbearing potential prior to starting the 50 Hz rTMS and also at the initial interview after signing the consent form. Women of childbearing potential will be asked to take appropriate measures to prevent a pregnancy during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aarsland D, Larsen JP, Waage O, Langeveld JH. Maintenance electroconvulsive therapy for Parkinson's disease. Convuls Ther. 1997 Dec;13(4):274-7. PMID 9437571
- [Background] Baudewig J, Siebner HR, Bestmann S, Tergau F, Tings T, Paulus W, Frahm J. Functional MRI of cortical activations induced by transcranial magnetic stimulation (TMS). Neuroreport. 2001 Nov 16;12(16):3543-8. doi: 10.1097/00001756-200111160-00034. PMID 11733708
- [Background] Belmaker RH, Grisaru N. Magnetic stimulation of the brain in animal depression models responsive to ECS. J ECT. 1998 Sep;14(3):194-205. PMID 9773358

RESULTS

PARTICIPANT FLOW:
Groups:
- Real rTMS: Subjects receiving real rTMS
- Sham rTMS: Subjects receiving sham rTMS.
Period: Overall Study
Arm/Group | Real rTMS | Sham rTMS
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real rTMS | Sham rTMS | Total
Number analyzed (Participants) | 13 | 13 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.1) | 63.7 (8.3) | 64.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 11 | 9 | 20
Duration of Disease [Mean (Standard Deviation); unit: years] | 8.6 (4.1) | 9.3 (6.8) | 8.96 (5.5)
Hoehn-Yahr, "on" [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The measurement on the Hoehn and Yahr was taken while the subject was on medication.
  units on a scale | 2.4 (0.2) | 2.5 (0.3) | 2.42 (.27)
Hoehn-Yahr "off" [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The measurement on the Hoehn and Yahr was taken while the subject was off medication.
  units on a scale | 2.7 (0.3) | 2.9 (0.6) | 2.8 (0.47)
Total LED [Mean (Standard Deviation); unit: milligrams] — Total levodopa-equivalent dose (medication) that subject is currently on
  milligrams | 861 (436) | 949 (677) | 905 (559.6)
Tremor [Number; unit: participants]
  Presence of Tremor | 10 | 12 | 22
  Absence of Tremor | 3 | 1 | 4
Gait freezing [Number; unit: participants]
  Presence of Gait Freezing | 7 | 9 | 16
  Absence of Gait Freezing | 6 | 4 | 10
Fluctuations [Number; unit: participants]
  Presence of Fluctuations | 7 | 8 | 15
  Absence of Fluctuations | 6 | 5 | 11
Dyskinesias [Number; unit: participants] — Presence or absence of dyskinesias (diminished voluntary movements and the presence of involuntary movements).
  participants
    Presence of dyskinesias | 4 | 5 | 9
    Absence of dyskinesias | 9 | 8 | 17
Falls [Number; unit: participants]
  Presence of falls | 1 | 0 | 1
  Absence of falls | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: Gait speed was assessed by measuring the time it takes to walk 10 meters. Subject's gait speed was measured while on medication and off medication for each group, i.e., real rTMS and sham rTMS. Two trials were averaged for each condition. Patients were instructed to walk fast without taking the risk of falling, wearing the same shoes and consistently using assistive devices if needed. Gait speed was measured at baseline and 1 day post intervention.
Time Frame: Baseline, 1 day post rTMS
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- On Medication Real rTMS: Subjects ON medication while receiving REAL rTMS
- On Medication Sham rTMS: Subjects ON medication while receiving SHAM rTMS
- Off Medication Real rTMS: Subjects OFF medication while receiving REAL rTMS
- Off Medication Sham rTMS: Subjects OFF medication while receiving SHAM rTMS
Arm/Group | On Medication Real rTMS | On Medication Sham rTMS | Off Medication Real rTMS | Off Medication Sham rTMS
Number analyzed (Participants) | 13 | 13 | 13 | 13
seconds
  Baseline | 7.54 (0.50) | 8.20 (0.50) | 8.31 (0.73) | 9.32 (0.76)
  1 day post rTMS | 6.89 (0.45) | 7.35 (0.45) | 7.41 (0.64) | 8.45 (0.67)

2. Secondary Outcome: Bradykinesia
Description: Bradykinesia refers to the slowness in executing a movement. Bradykinesia was assessed by measuring the time in seconds it takes to do the following sequence, 10 times: 1) hand closing and opening while squeezing a ball 2) elbow flexion 3) hand closing and opening, and 4) elbow extension. Subjects were allowed to practice these hand and arm movements until performance appeared not to get faster, and then abstained from further practice to minimize learning effects. The time it takes subjects to execute the entire sequence 10 times with either the left or right arm/hand was measured. Means are reported for each group.
Time Frame: Baseline, 1 day post rTMS
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- On Medictation Sham rTMS: Subjects ON medication while receiving SHAM rTMS
Arm/Group | On Medication Real rTMS | On Medictation Sham rTMS | Off Medication Real rTMS | Off Medication Sham rTMS
Number analyzed (Participants) | 13 | 13 | 13 | 13
seconds
  Baseline | 12.86 (0.71) | 11.46 (0.74) | 14.12 (0.86) | 12.90 (0.93)
  1 day post rTMS | 10.17 (0.65) | 9.30 (0.68) | 10.48 (0.62) | 9.65 (0.67)

3. Secondary Outcome: Total UPDRS Score
Description: The Total Unified Parkinson's Disease Rating Scale (UPDRS) is an overall assessment scale that quantifies the signs and symptoms of Parkinson's disease. The total UPDRS score consists of mentation, behavior, mood, activities of daily living and motor components, and ranges from 0 (not affected) to 176 (most severely affected). The total UPDRS score is obtained from patient examination, interview and patient questionnaires.
Time Frame: Baseline, 1 day post rTMS
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Medication Real rTMS | On Medictation Sham rTMS | Off Medication Real rTMS | Off Medication Sham rTMS
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale
  Baseline | 49.31 (4.1) | 48.92 (4.3) | 57.77 (4.2) | 58.75 (4.2)
  1 day post rTMS | 45.00 (4.2) | 47.67 (4.4) | 53.46 (4.0) | 57.75 (4.2)

4. Secondary Outcome: Motor UPDRS
Description: The Motor Unified Parkinson's Disease Rating Scale (UPDRS) includes only the motor assessment of the UPDRS (Part III) and examines speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability and body bradykinesia. The scores range from 0 (no motor impairment) to 108 (severe motor impairment). The Motor UPDRS was administered at baseline and at 1 day post rTMS or sham. Subjects were assessed on medication and off medication.
Time Frame: Baseline, 1 day post rTMS
Population: Intent to treat.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Off Medictation Real rTMS: Subjects OFF medication while receiving REAL rTMS
Arm/Group | On Medication Real rTMS | Off Medictation Real rTMS | On Medication Sham rTMS | Off Medication Sham rTMS
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale
  Baseline | 32.08 (2.5) | 30.00 (2.6) | 38.46 (2.2) | 37.25 (2.3)
  1 day post rTMS | 29.85 (2.7) | 29.58 (2.8) | 36.46 (2.3) | 36.50 (2.4)

5. Secondary Outcome: Activities of Daily Living UPDRS
Description: The Activities of Daily Living Unified Parkinson's Disease Rating Scale (ADL UPDRS) is a self evaluation of the activities of daily living. The following variables are rated: speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed, falling, freezing when walking, walking, tremor and sensory complaints. Each variable is rated on a scale of 0 (normal) to 4 (severe impairment). A total score for the ADL UPDRS ranges from 0 (no impairment) to 52 (severe impairment).
Time Frame: Baseline, 1 day post rTMS
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Medication Real rTMS | On Medictation Sham rTMS | Off Medication Real rTMS | Off Medication Sham rTMS
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale
  Baseline | 11.15 (1.3) | 12.58 (1.4) | 13.23 (1.5) | 15.17 (1.6)
  1 day post rTMS | 9.39 (1.4) | 11.33 (1.5) | 11.23 (1.6) | 14.50 (1.7)

ADVERSE EVENTS:
Arm/Group | On Medication Real rTMS | Off Medictation Real rTMS | On Medication Sham rTMS | Off Medication Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes